CLINICAL TRIAL: NCT05879276
Title: Effect at 3 Months of Early Empagliflozin Initiation in Cardiogenic Shock Patients on Mortality, Rehospitalization, Left Ventricular Ejection Fraction and Renal Function. A Randomized Multicentric Open Trial
Brief Title: Effect at 3 Months of Early Empagliflozin Initiation in Cardiogenic Shock Patients on Mortality, Rehospitalization, Left Ventricular Ejection Fraction and Renal Function.
Acronym: EMPASHOCK
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Dr Antoine KIMMOUN, coordinating investigator, Central Hospital, Nancy, France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023PI223 - 2023-503602-37-00
Record Dates: First submitted 2023-04-12; First posted 2023-05-30 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Cardiogenic Shock
Keywords: Heart failure; Acute heart failure; Cardiogenic shock; SGLT2 inhibitor; Mortality
MeSH Terms: conditions — Shock, Cardiogenic; Heart Failure | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Multicentre, interregional, randomised, controlled, open-label clinical trial evaluating the effect of early initiation of a SGLT2 inhibitor i.e Empaglifozin, in cardiogenic shock.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empaglifozin in addition to standard management (Experimental): Patients in cardiogenic shock receiving empagliflozin in addition to standard management at a dose of 10 mg per day per os (or through nasogastric tube in intubated patients) for a duration of 12 weeks
  Interventions: Drug: Empagliflozin 10 MG
- Standard management (No Intervention): Patients in cardiogenic shock receiving a standard management. SGLT2 inhibitor, which are now standard of care in chronic heart failure, in the strict respect of their indications, could be prescribed in the standard management group after hospitalization discharge.

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Patients in cardiogenic shock receiving empagliflozin in addition to standard management at a dose of 10 mg per day per os (or through nasogastric tube in intubated patients) for a duration of 12 weeks.
  Arms: Empaglifozin in addition to standard management

SUMMARY:
Long term prognosis of cardiogenic shock is related to the resolution of haemodynamic failure, associated visceral failure and the recovery of an adequate myocardial function. In the immediate aftermath of cardiogenic shock, after catecholamines weaning, there are no recommendations on cardiovascular treatments that would improve this long term prognosis. Indeed, the standard cardiovascular treatments such as inhibitors of the renin-angiotensin and aldosterone system and beta-blockers have hypotensive and negative inotropic effects and may worsen the renal function. In practice, given their side effects, they are not prescribed in the immediate aftermath of cardiogenic shock.

Sodium-glucose co-transporter 2 (iSGLT2) inhibitors are now an integral part of the drug management of chronic heart failure and the EMPULSE-HF trial has just demonstrated a benefit in acute heart failure (PMID: 35228754). Several pivotal clinical trials have demonstrated a significant effect of iSGLT2 on the survival and the risk of re hospitalisation for heart failure (PMID: 32865377, 31535829, 33200892). Our hypothesis is that, in patients in cardiogenic shock, early treatment with Empaglifozin in addition to the standard management could reduce mortality and morbidity (death, transplantation/LVAD and rehospitalisation for heart failure) and improve myocardial function at 12 weeks, compared with standard management alone.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients hospitalized in critical cardiac unit care or Intensive care unit for a cardiogenic shock
* "Who must have been or is on catecholamines for at least 12 hours for the treatment of cardiogenic shock.
* Patients who are able to take oral tablets

Exclusion Criteria:

* GFR< 20 ml/min/1.73m2.
* Chronic dialysis.
* Patient on SGLT2 inhibitors prior to admission to ICU or CCU.
* Known allergy to SGLT2 inhibitors or to any of its excipients (in particular, patients with hereditary disorders of galactose intolerance, total lactase deficiency or glucose or galactose malabsorption syndrome)
* Patients on lithium.
* Patient in shock for another cause or moribund (SAPS2> 90).
* Specific cardiogenic shock context:

  1. cardiac transplant patient or on transplant list.
  2. peripartum, adrenergic, valvular, non ischemic, post embolic heart disease.
  3. related to cardiotropic drug intoxication.
  4. Secondary to a cardiac arrest for which the patient remains comatose prior to inclusion.
* Women of childbearing age without effective contraception.
* Person referred to in Articles 10, 31, 32, 33 and 34 of EU Regulation 536/2014 (Pregnant woman, parturient or breastfeeding mother, Minor (not emancipated), Adult person subject to a legal protection measure (guardianship, curatorship, safeguard of justice))

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2027-03-16 (Estimated); Study Completion 2027-03-16 (Estimated)

PRIMARY OUTCOMES:
Time to all-cause death | 12-week after randomisation
  To compare the effect of early introduction of empagliflozin in addition to standard management versus standard management alone on composite endpoint components:
  1. All-cause mortality or heart transplantation or ventricular assist,
  2. Rehospitalization for heart failure,
  3. Left ventricular ejection fraction.
  Hierarchical composite endpoint, assessed at 12 weeks from randomization (win-ratio method):
  * Rank 1: Time to all-cause death or cardiac transplantation or mechanical ventricular assist,
  * Rank 2: Time to rehospitalization for heart failure,
  * Rank 3: Left ventricular ejection fraction assessed during a research cardiac ultrasound.
Time to cardiac transplantation | 12-week after randomisation
  To compare the effect of early introduction of empagliflozin in addition to standard management versus standard management alone on composite endpoint components:
  1. All-cause mortality or heart transplantation or ventricular assist,
  2. Rehospitalization for heart failure,
  3. Left ventricular ejection fraction.
  Hierarchical composite endpoint, assessed at 12 weeks from randomization (win-ratio method):
  * Rank 1: Time to all-cause death or cardiac transplantation or mechanical ventricular assist,
  * Rank 2: Time to rehospitalization for heart failure,
  * Rank 3: Left ventricular ejection fraction assessed during a research cardiac ultrasound.
Time to mechanical ventricular assist | 12-week after randomisation
  To compare the effect of early introduction of empagliflozin in addition to standard management versus standard management alone on composite endpoint components:
  1. All-cause mortality or heart transplantation or ventricular assist,
  2. Rehospitalization for heart failure,
  3. Left ventricular ejection fraction.
  Hierarchical composite endpoint, assessed at 12 weeks from randomization (win-ratio method):
  * Rank 1: Time to all-cause death or cardiac transplantation or mechanical ventricular assist,
  * Rank 2: Time to rehospitalization for heart failure,
  * Rank 3: Left ventricular ejection fraction assessed during a research cardiac ultrasound.
Time to rehospitalization for heart failure. | 12-week after randomisation
  To compare the effect of early introduction of empagliflozin in addition to standard management versus standard management alone on composite endpoint components:
  1. All-cause mortality or heart transplantation or ventricular assist,
  2. Rehospitalization for heart failure,
  3. Left ventricular ejection fraction.
  Hierarchical composite endpoint, assessed at 12 weeks from randomization (win-ratio method):
  * Rank 1: Time to all-cause death or cardiac transplantation or mechanical ventricular assist,
  * Rank 2: Time to rehospitalization for heart failure,
  * Rank 3: Left ventricular ejection fraction assessed during a research cardiac ultrasound.
Left ventricular ejection fraction assessed by cardiac ultrasound. | 12-week after randomisation
  To compare the effect of early introduction of empagliflozin in addition to standard management versus standard management alone on composite endpoint components:
  1. All-cause mortality or heart transplantation or ventricular assist,
  2. Rehospitalization for heart failure,
  3. Left ventricular ejection fraction.
  Hierarchical composite endpoint, assessed at 12 weeks from randomization (win-ratio method):
  * Rank 1: Time to all-cause death or cardiac transplantation or mechanical ventricular assist,
  * Rank 2: Time to rehospitalization for heart failure,
  * Rank 3: Left ventricular ejection fraction assessed during a research cardiac ultrasound.

SECONDARY OUTCOMES:
Death | 12-week after randomisation
  To compare the effect of early introduction of empagliflozin in addition to standard management versus standard management alone on all-cause mortality at 12 weeks from randomization
Heart transplantation or long-term ventricular assistance | 12-week after randomisation
  To compare the effect of early introduction of empagliflozin in addition to standard management versus standard management alone on heart transplantation or long-term ventricular assistance, at 12 weeks from randomization
Rehospitalization for heart failure | from hospital discharge to 12-week after randomisation
  To compare the effect of early introduction of empagliflozin in addition to standard management versus standard management alone on rehospitalization for heart failure, at 12 weeks from randomization
Left ventricular ejection fraction assessed by cardiac ultrasound. | 12-week after randomisation
  To compare the effect of early introduction of empagliflozin in addition to standard management versus standard management alone on left ventricular ejection fraction, at 12 weeks from randomization.
E' wave assessed by cardiac ultrasound | 12-week after randomisation
  To compare the effect of early introduction of empagliflozin in addition to standard management versus standard management alone on the left ventricular diastolic function and filling pressures, at 12 weeks from randomization.
E/e' ratio assessed by cardiac ultrasound | 12-week after randomisation
  To compare the effect of early introduction of empagliflozin in addition to standard management versus standard management alone on the left ventricular diastolic function and filling pressures, at 12 weeks from randomization.
TAPSE assessed by cardiac ultrasound | 12-week after randomisation
  To compare the effect of early introduction of empagliflozin in addition to standard management versus standard management alone on the right ventricular function, at 12 weeks from randomization
S wave at the annular tricuspid level assessed by cardiac ultrasound | 12-week after randomisation
  To compare the effect of early introduction of empagliflozin in addition to standard management versus standard management alone on the right ventricular function, at 12 weeks from randomization
Renal replacement therapy | Randomisation and 12-week after randomisation
  To compare the effect of early introduction of empagliflozin in addition to standard management versus standard management alone on the renal function, at 12 weeks from randomization
Renal function | Randomisation and 12-week after randomisation
  The number of patients requiring renal replacement therapy between randomization and 12 weeks, and change in renal function assessed at baseline and 12 weeks: glomerular filtration rate calculated by the CKD-EPI method
Bilirubin | Randomisation and 12-week after randomisation
  To compare the effect of early introduction of empagliflozin in addition to standard management versus standard management alone on the hepatic function, at 12 weeks from randomization
Prothrombin Ratio (PT) | Randomisation and 12-week after randomisation
  To compare the effect of early introduction of empagliflozin in addition to standard management versus standard management alone on the hepatic function, at 12 weeks from randomization
SGOT | Randomisation and 12-week after randomisation
  To compare the effect of early introduction of empagliflozin in addition to standard management versus standard management alone on the hepatic function, at 12 weeks from randomization
SGPT | Randomisation and 12-week after randomisation
  To compare the effect of early introduction of empagliflozin in addition to standard management versus standard management alone on the hepatic function, at 12 weeks from randomization
NT-Pro-BNP | Randomisation and 12-week after randomisation
  To compare the effect of early introduction of empagliflozin in addition to standard management versus standard management alone on the evolution of the hydro-sodic overload, at 12 weeks from randomization. The measure of NT-Pro-BNP will be measured at 12 weeks and delta from randomisation will be calculated
Weight | Randomisation and 12-week after randomisation
  To compare the effect of early introduction of empagliflozin in addition to standard management versus standard management alone on the evolution of the hydro-sodic overload, at 12 weeks from randomization. The weight will be measured at 12 weeks and delta from randomisation will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas GIRERD, MD PhD, Study Chair — CHRU of NANCY
Locations (8):
- France (8):
  - CHR Metz - Thionville, Ars-Laquenexy
  - CHU de Besançon, Besançon
  - CHU de Dijon Bourgogne, Dijon
  - CHU Lille, Lille
  - CHU Reims, Reims
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHRU de NANCY - réanimation médicale, Vandœuvre-lès-Nancy
  - Chru Nancy - Usic, Vandœuvre-lès-Nancy